CLINICAL TRIAL: NCT01208415
Title: PRESERVE-Zenith® Iliac Branch System Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-625-P1
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2017-09

CONDITIONS: Aorto-iliac Aneurysms; Iliac Aneurysms
Keywords: Zenith aortoiliac aneurysm; iliac aneurysm; branch; connections; endovascular graft; graft-iliac bifurcation; Aneurysm; Vascular Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Iliac Aneurysm; Aneurysm; Vascular Diseases; Cardiovascular Diseases

ARMS (1):
- Device Implant (Experimental)
  Interventions: Device: Endovascular repair for aortoiliac or iliac aneurysms.

INTERVENTIONS:
Device: Endovascular repair for aortoiliac or iliac aneurysms. — Implantation of the Zenith® Branch Endovascular Graft-Iliac Bifurcation, the Zenith® Connection Endovascular Covered Stent/ConnectSX™ and the Zenith® Flex AAA Endovascular Graft.
  Other Names: Endovascular repair for aortoiliac or iliac aneurysm.

SUMMARY:
The PRESERVE-Zenith® Iliac Branch System Clinical Study is a clinical trial to study the safety and effectiveness of the Zenith® Branch Endovascular Graft-Iliac Bifurcation in combination with the Zenith® Connection Endovascular Stent/ConnectSX™ covered stent in the treatment of aorto-iliac and iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* An aortoiliac or iliac aneurysm of appropriate size
* Unsuitable distal sealing site for a traditional Zenith® iliac leg graft within the common iliac artery

Exclusion Criteria:

* Less than 18 years of age
* Inability or refusal to give informed consent
* Disease considerations that would compromise patient safety or study outcomes
* Unsuitable arterial anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2017-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Anthony Lee, MD, FACS, Principal Investigator — Christine E. Lynn Heart and Vascular Institute
Locations (19):
- United States (19):
  - VA Palo Alto HCS, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - Christine E. Lynn Heart and Vascular Institute, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Massachusetts, Worcester, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital East Communities, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
  - Aurora St. Luke's Hospital, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Zenith® Iliac Branch System: Zenith® Branch Endovascular Graft-Iliac Bifurcation System is made up of two devices: the Zenith® Branch Endovascular Graft-Iliac Bifurcation and the ConnectSX™.
Period: Overall Study
Arm/Group | Zenith® Iliac Branch System
Started | 40
6 Months | 37
Completed | 0
Not Completed | 40
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Device not placed | 1
Not completed — Still be eligible for follow-up | 33

BASELINE CHARACTERISTICS:
Arm/Group | Zenith® Iliac Branch System
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Patients That Are Free From Patency-related Intervention
Description: Patency-related intervention is defined as: Secondary intervention to treat a > 60% stenosis of the internal iliac artery (as identified through CT, angiography, or duplex ultrasound and confirmed by core laboratory) associated with clinical symptoms. Of note, this not only includes patients with internal iliac artery stenosis following successful placement of the Zenith® Branch Endovascular Graft-Iliac Bifurcation and ConnectSX™, but also any cases of technical failure resulting in occlusion of the internal iliac artery during the initial implant procedure that require secondary intervention for associated clinical symptoms.
Time Frame: 6 Months
Population: Of the 37 patients available for analysis at 6 months, data was available for 34 patients.
Measure: Number; unit: participants
Arm/Group | Device Implant
Number analyzed (Participants) | 34
participants | 33

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Zenith® Iliac Branch System
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 7/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Iliac Branch System (N=40)
Hypotension (Cardiac disorders) | 1 (1)
Spinal cord infarct (Nervous system disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Confusion (General disorders) | 1 (1)
Non-Hodgkins lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bursitis with overlying cellulitis (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Iliac Branch System (N=40)
Groin seroma (Surgical and medical procedures) | 3 (3)
Groin hematoma (Surgical and medical procedures) | 2 (2)
Urinary retention (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days